CLINICAL TRIAL: NCT02226770
Title: Heart-focused Anxiety in Patients With Implantable Cardioverter Defibrillator (ICD) and/or Mechanical Cardiovascular Assist Device (AD) (Anxiety-CHF)
Brief Title: Heart-focused Anxiety in Patients With Heart Failure and ICD
Acronym: Anxiety-CHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Collaborators: Friede Springer Herz Stiftung (Unknown)
Responsible Party: Principal Investigator, Ingird Kindermann (PD Dr. med), Prof. Dr. med., University Hospital, Saarland
Organization: Universität des Saarlandes (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 252/12
Record Dates: First submitted 2014-04-17; First posted 2014-08-27 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure Patients Before and After ICD Implantation
MeSH Terms: interventions — Defibrillators, Implantable

ARMS (1):
- ICD (Other): Implantation of an Implantable Cardioverter Defibrillator (ICD) in patients with heart failure
  Interventions: Device: Implantable Cardioverter Defibrillator (ICD)

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator (ICD)

SUMMARY:
The aim of the present study is to measure heart-focused anxiety, general anxiety, depression, PTSD and quality of life as well as type D personality in patients with heart failure before and after the implantation of a cardioverter defibrillator (ICD) and/or assist device (AD).

DETAILED DESCRIPTION:
In patients with heart failure and implantable Cardioverter Defibrillator (ICD) psychological comorbidities such as heart focused anxiety and depression often occur. These psychological factors may have negative effects on compliance as well as on the development of the cardiac disease and therefore on rehospitalization and mortality rates.

A personality structure where negative affect is paired with social inhibition (the inability to communicate ones feelings to others) can often be found in patients with cardiovascular disease. This so-called type D personality is also associated with a worse prognosis.

It is of interest whether, and if so in what way, the implantation of an ICD can affect the psychological well-being and through that the prognosis of the heart failure patient.

The goal of this study is therefore to investigate the effect of ICD implantation on heart-focused anxiety, depression, possible traumatization and quality of life in patients with heart failure with consideration of a possible moderating effect of the type D personality.

Furthermore, the impact of the above stated psychological factors on rehospitalization and mortality, as well as on frequency of shocks shall be examined.

Vice versa, the frequency of shocks or the impact of being shocked at all on psychological factors is of interest.

ELIGIBILITY:
Inclusion Criteria:

* heart failure, indication for an implantable Cardioverter Defibrillator

Exclusion Criteria:

* psychosis; advanced dementia; drug abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2010-07-14 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2016-10-28 (Actual)

PRIMARY OUTCOMES:
Extent of heart-focused anxiety before and change after ICD implantation | From baseline before ICD implantation to 24 months after implantation
  Heart-focused anxiety is measured through the use of the Cardiac Anxiety Questionnaire. All questionnaires will be filled out at baseline (before device implantation) as well as 5, 12 and 24 months after implantation.
Extent of general anxiety and depression before and change after ICD implantation | From baseline before ICD implantation to 24 months after implantation
  General anxiety and depression are recorded with the Hospital Anxiety and Depression Scale.
  All questionnaires will be filled out at baseline (before device implantation) as well as 5, 12 and 24 months after implantation.
Quality of life before and change after ICD implantation | From baseline before ICD implantation to 24 months after implantation
  Quality of life is documented through the Minnesota Living With Heart Failure Questionnaire.
  All questionnaires will be filled out at baseline (before device implantation) as well as 5, 12 and 24 months after implantation.
Number of patients affected by PTSD before and after ICD implantation | From baseline before ICD implantation to 24 months after implantation
  The Impact of Event Scale (revised) is used to evaluate the possibility of a post-traumatic stress disorder (PTSD).
  All questionnaires will be filled out at baseline (before device implantation) as well as 5, 12 and 24 months after implantation.

SECONDARY OUTCOMES:
Impact of type D personality on heart-focused anxiety | For type D: Baseline and for the psychological variable: from baseline before ICD implantation to 24 months after implantation
  Type D ist measured with the Type D Scale-14 (DS14). Heart-focused anxiety is measured as stated in the primary outcome measures section.
Impact of type D personality on general anxiety and depression | For type D: Baseline and for the psychological variables: from baseline before ICD implantation to 24 months after implantation.
  Type D ist measured with the DS14. General anxiety and depression are measured as stated in the primary outcome measures section.
Impact of type D personality on quality of life. | For type D: Baseline and for the psychological variable: from baseline before ICD implantation to 24 months after implantation.
  Type D ist measured with the DS14. Quality of life is measured as stated in the primary outcome measures section.
Impact of type D personality on PTSD. | For type D: Baseline and for the psychological variable: from baseline before ICD implantation to 24 months after implantation.
  Type D ist measured with the DS14. PTSD is measured as stated in the primary outcome measures section.
Impact of type D personality on numbers of shocks. | For type D: Baseline and for number of shocks: from ICD implantation to 24 months after implantation.
  Type D ist measured with the DS14. ICD-shocks will be measured as number of shocks per patient.
Impact of type D Personality on rehospitalization and morbidity. | For type D: Baseline and for rehospitalization and morbidity: from implantation until 24 months after implantation..
  Type D ist measured with the DS14. Psychological factors will be measured as stated in the primary outcomes section.
  Rehospitalization will be measured as number of times of readmission and mortality will be measured in total numbers of patients.
Influence of heart-focused anxiety on rehospitalization and morbidity | Baseline to 24 months after implantation.
  Heart-focused anxiety will be measured as stated in the primary outcomes section.
  Rehospitalization will be measured as number of times of readmission and mortality will be measured in total numbers of patients.
Influence of general anxiety and depression in rehospitalization and morbidity | Baseline to 24 months after implantation.
  General anxiety and depression will be measured as stated in the primary outcomes section.
  Rehospitalization will be measured as number of times of readmission and mortality will be measured in total numbers of patients.
Influence of quality of life on rehospitalization and morbidity | Baseline to 24 months after implantation.
  Quality of life will be measured as stated in the primary outcomes section. Rehospitalization will be measured as number of times of readmission and mortality will be measured in total numbers of patients.
Effect of ICD-shocks on heart-focused anxiety and effect of heart-focused anxiety on frequency of shocks | Baseline to 24 months after implantation.
  Heart-focused anxiety will be measured as stated in the primary outcomes section.
  ICD-shocks will be measured as number of shocks per patient.
Effect of ICD-shocks on general anxiety and depression and effect of general anxiety and depression on frequency of shocks | Baseline to 24 months after implantation.
  General anxiety and depression will be measured as stated in the primary outcomes section.
  ICD-shocks will be measured as number of shocks per patient.
Effect of ICD-shocks on quality of life and effect of quality of life on frequency of shocks | Baseline to 24 months after implantation.
  Quality of life will be measured as stated in the primary outcomes section. ICD-shocks will be measured as number of shocks per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Kindermann, PD Dr. med., Principal Investigator — Saarland University Hospital; Denise Lenski, Dr. rer. nat. Dipl.-Psych., Principal Investigator — Saarland University Hospital; Maxie Bunz, Dipl.-Psych., Principal Investigator — Saarland University Hospital
Locations (1):
- Saarland University Hospital, Homburg, Saarland, Germany

REFERENCES:
- [Derived] Bunz M, Lenski D, Wedegartner S, Ukena C, Karbach J, Bohm M, Kindermann I. Heart-focused anxiety in patients with chronic heart failure before implantation of an implantable cardioverter defibrillator: baseline findings of the Anxiety-CHF Study. Clin Res Cardiol. 2016 Mar;105(3):216-24. doi: 10.1007/s00392-015-0909-1. Epub 2015 Oct 19. PMID 26481915